CLINICAL TRIAL: NCT02110979
Title: Validation of a Patient Decision Aid for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EPI-Q (Other)
Responsible Party: Principal Investigator, Alicia Shillington, Executive Vice President, EPI-Q
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 70-1036-015
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Patient Decision Aid; Shared Decision Making
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDA (Experimental): Subjects receive an internet-based patient decision aid video. The PDA is viewed outside of the doctor's office via a personal computer in preparation for regularly scheduled face to face interaction between patients and clinicians.
  Interventions: Behavioral: Use of a PDA to assist shared decision making
- Usual care (No Intervention): Patients receive usual care as determined by their clinician.

INTERVENTIONS:
Behavioral: Use of a PDA to assist shared decision making
  Other Names: Patient Decision Aid
  Arms: PDA

SUMMARY:
The objectives of this study are to compare measurements in knowledge of decision options, support for decision making, uncertainly in decision making, and clarity of values important to decision making among two groups of type 2 diabetes patients, those who receive a Patient Decision Aid and those who receive usual care.

DETAILED DESCRIPTION:
This study uses a randomized, controlled trial design to compare knowledge of decision options, support for decision making, uncertainly in decision making, and clarity of values important to decision making among patients with uncontrolled type 2 diabetes who are only taking metformin medication. The intervention is a Patient Decision Aid (PDA) video delivered via the internet.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Age 18 or older
3. English speaking
4. Currently taking metformin
5. Inadequate glycemic control in the opinion of the investigator
6. Is considering additional medication options on the advice of their physician
7. Can provide a valid email address
8. Access to the internet and able to read and respond to internet questionnaires

Exclusion Criteria:

1. Participation in a clinical trial of a diabetes medication within 1 year
2. Currently taking more than two (2) medications for diabetes
3. Has been exposed to diabetes medications from more than three (3) drug classes
4. Adults unable to consent
5. Individuals who are not yet adults (infants, children, teenagers)
6. Pregnant women
7. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Knowledge score | 6 weeks
  The primary endpoint for this investigation is the knowledge total score at final followup 4- 6 weeks after randomization between the PDA versus usual care groups. Questions are about available treatments and specific to the information on medication options available to people with type 2 diabetes when metformin alone does not achieve adequate glycemic control.

SECONDARY OUTCOMES:
Decisional conflict | 6 weeks
  Measured by using the Decisional Conflict Scale (DCS). Scale will measure domains including: (1) uncertainty in choosing among alternatives; (2) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about values and unsupported in decision making; and (3) perceived quality of decision making. Global decision conflict score and perceived effective decision sub-score will be summarized descriptively following decision and will be compared between arms. Sub-scores are: Uncertainty, Informed, Values clarity, and Support.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Shillington, PhD, Principal Investigator — EPI-Q
Locations (2):
- United States (2):
  - EPI-Q Inc, Oak Brook, Illinois
  - EPI-Q, Oak Brook, Illinois

REFERENCES:
- [Derived] Bailey RA, Pfeifer M, Shillington AC, Harshaw Q, Funnell MM, VanWingen J, Col N. Effect of a patient decision aid (PDA) for type 2 diabetes on knowledge, decisional self-efficacy, and decisional conflict. BMC Health Serv Res. 2016 Jan 14;16:10. doi: 10.1186/s12913-016-1262-4. PMID 26762150